CLINICAL TRIAL: NCT01078064
Title: Gastric Accommodation as a Factor Influencing the Number of Reflux Episodes in Children and Adolescents
Brief Title: Gastric Accommodation and Gastroesophageal Reflux
Status: Terminated | Type: Observational
Why Stopped: the study failed in recruiting the required number of subjects (sample size) during its period
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Rodrigo Strehl Machado, MD, PhD, Nationwide Children's Hospital
Other Study IDs: 001-2010
Record Dates: First submitted 2010-02-25; First posted 2010-03-02 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal reflux disease, gastric motility
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: Patients with symptoms suggesting gastroesophageal reflux and referred to perform an impedance study.

SUMMARY:
Gastroesophageal reflux events generally happen during relaxation of lower esophageal sphincter. This relaxation is a reflex that is triggered by gastric stimuli. The investigators hypothesize that abnormal relaxation of the gastric wall after a meal may lead to reflux events. To test this hypothesis, a study was designed to measure the gastric accommodation in patients undergoing esophageal impedance monitoring.

DETAILED DESCRIPTION:
Gastroesophageal reflux events happen during relaxations of lower esophageal sphincter not related to swallowing, called transient. These transient lower esophageal sphincter relaxations (tLESR) are generally triggered by gastric distension and its physiological purpose is to vent the stomach. The gastric accommodation is a physiological process in which the gastric fundus actively relaxes during a meal in order to accommodate it.

This study is driven by the hypothesis that impairment of the gastric accommodation may facilitate triggering tLESR and, therefore, reflux events. We aim to evaluate the relation between gastric fundic relaxation and the number of gastroesophageal reflux events in children. We also aim to evaluate if there is a relation between the gastric emptying and the number of reflux episodes.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents older than 1-year old who were referred for combined esophageal impedance pH monitoring for GERD* symptoms

Exclusion Criteria:

* continuous feeding
* previous fundoplication

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children and adolescents older than 1-year old who were referred for combined esophageal impedance pH monitoring for GERD symptoms, such as epigastric pain, respiratory symptoms, heartburn, feeding difficulties, chest pain, nausea or vomiting.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
NUMBER OF REFLUX EPISODES | 1 day
  It is a cross-sectional exam, and the number of reflux episodes at baseline, after a clinically indicated 24-hour impedance study

SECONDARY OUTCOMES:
Gastric volume ratio: 10 min/baseline | 1 day
  It is a cross-sectional study. This variable will be assessed by ultrasound in the next morning of the impedance study.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo S Machado, MD, PhD, Principal Investigator — Nationwide Children's Hospital; Beth Skaggs, CCRC, Study Director — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States